CLINICAL TRIAL: NCT04595656
Title: Defining Burden of Diseases and Causes of Deaths Using Electronic Verbal Autopsy Methods in Rural South and Southeast Asia: A Multi-centre Study in Bangladesh, Lao PDR, and Myanmar
Brief Title: Defining Causes of Deaths in South and Southeast Asia
Acronym: SEACTN-VA
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: HCR20007
Record Dates: First submitted 2020-10-12; First posted 2020-10-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cause of Mortality; Cause of Neonatal Death; Cause of Child Death; Cause of Maternal Death; Cause of Adult Death
Keywords: Death; fatal outcome; interview; mortality; pathologic process
MeSH Terms: conditions — Death; Pathologic Processes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: verbal autopsy interview — The study involves filling of verbal autopsies for deaths in SEACTN villages. This is an observational study being conducted as a substudy of rural febrile project of SEACTN program.

SUMMARY:
Mortality data are important in low and middle-income countries to assess the population health status and trends. Mortality statistics in the populations of Bangladesh, Myanmar and Lao PDR are considered as generally limited and a recent assessment of vital registration systems of those countries reported a poor performance of the death registration system. Majority of deaths occur at home in rural area of those countries without cause of death assigned. To address this problem, the investigators will use verbal autopsy (VA) method developed by WHO to ascertain the cause of a death based on an interview with a family member or caregiver of deceased person to obtain information about causes of death in study rural communities. Death related to a specific cause will be defined by ICD-10 codes and described as primary, secondary or underlying COD. The study is planned to conduct in approximately 390 rural village communities covered by Southeast Asia clinical trial network (SEACTN) network in proposed 3 countries. The study findings will help establish a better understanding in signs, symptoms, medical history and circumstances preceding death; prioritize future interventions for early and effective diagnostics and treatment for diseases and how to keep mortality surveillance ongoing in study rural settings.

DETAILED DESCRIPTION:
The SEACTN (South and Southeast Asian Community-based Trials Network) is a part of a portfolio of programmes under the Wellcome Innovations Flagship 'Innovations for Impact in Resource-limited Settings'. The flagship plan is to build the SEACTN infrastructure in approximately 520 villages across three South and Southeast Asian countries (Bangladesh, Lao PDR and Myanmar) to capture over 100,000 episodes and outcomes of rural febrile illness in these remote and underserved communities. Mortality statistics in the populations covered by SEACTN are considered as generally limited and unreliable and a recent assessment of vital registration systems of these 3 countries showed a poor performance of the death registration system. To support the goal of the flagship SEACTN program in defining the morbidity and mortality burden of febrile illness and to strengthen the mortality data (causes of deaths information) in study areas, the VA component is integrated as a part of project activities. It will identify not only potential causes of deaths with a history of febrile illnesses, but also all other CODs which occur in SEACTN network communities. The findings will also uncover large gaps and challenges that impede delivery of primary health services in rural area of the countries.

This observational multicountry study aims to conduct verbal autopsies in approximately 390 rural village communities in the SEACTN network in 5 countries; Bangladesh (in Cox's Bazar and Bandarban districts), Lao PDR (in Phalanxay, Phin and Atsaphanthong districts in the Province of Savannakhet), Thailand (Muang district of Chiang Rai province), Cambodia (Battambang and Pailin provinces)and Thai-Myanmar border area (Kayin state, Myanmar). The study populations are restricted to varying degrees from accessing adequate health services due to geographical and financial factors. Since VA interviews will be carried out for all deaths, the study will be able to point out capacity gaps in providing essential health services at different levels of the health system as well as barriers in receiving healthcare services. About 2,000 deaths or VA interviews are expected to be carried out over a 2-year study period.

Study procedure: The death cases in villages will be notified by village health workers (VHWs) or community health workers (CHWs) and also be checked through health facilities records. The study respondent should be a close family member or a caregiver or a person who closely attended to the deceased during the illness. VA instrument Questionnaires WHO 2016 version of validated electronic VA questionnaires will be used and there are three separate VA forms for specific age groups: perinatal and neonatal mortality (death of a child under 4 weeks), child mortality (aged 4 weeks to 11 years), adult mortality (aged 12 years and over) including maternal mortality. VA cause of death list The WHO VA cause of death list is used to classify disease. The COD list is based on the international classification of diseases (ICD-10) coding system.

The training of interviewers will be via online and face to face training sessions. The training materials from research collaborators (University of Toronto, Canada) will be used and adapted in local context. There will also be web based intensive courses for physicians for coding and CoD certification. A VA needs an optimum recall period for high quality of information. To keep the recall period as short as possible and to get reliable information, field team will aim to visit the villages at 3-6 months intervals and conduct interviews with the respondents of deceased persons to collect the information. The interview will take approximately 30 to 45 minutes to complete using electronic format of questionnaires installed in CommCare apps of SEACTN tablets after getting informed consent. Audio recordings will be done to make sure for accurate records of the interviews and to complete the narrative text section of the form. The investigators will also record the location of the villages by GPS in order to define causes of deaths with a map.

For quality control of the interview process, 10 percent of interviews will be observed and checked by field supervisors while conducting interviews. For quality control of coding and, assessing the COD, two physicians will independently review the outcome of an interview, will provide coding and formulate a COD. The COD identified by each physician will be recorded in the database and if there is any disagreement, a third senior physician would be brought in to adjudicate the result and sought for a solution.

ELIGIBILITY:
Inclusion Criteria:

* All adult participants whose family member's death occurred in SEACTN villages within 12 months.

Exclusion Criteria:

* Participants whose family member's death occurred outside of SEACTN villages or deaths more than 12months
* Respondents who are not providing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The respondent should be a close family member or a caregiver or a person who closely attended to the deceased during the illness (e.g. the mother in the case of an infant death, the spouse in case of an adult death, the son/daughter in the case of deaths among the elderly and an adult female relative in case of maternal deaths); and the respondent's educational status and communication skills. If needed, another household member or neighbor can help the primary respondents for specific details.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
~2,000 deaths classified according to ICD-10 classification | 18-20 months recruitment
  Classification of causes of deaths by verbal autopsy methods in rural areas of South and Southeast Asia: Based on information from the VA interview, the study physicians will identify possible causes of death. Death related to a specific cause will be defined by ICD-10 codes and described as primary, secondary or underlying COD.

SECONDARY OUTCOMES:
Age standardized mortality rate, gender specific CODs | 18-20 months of recruitment period
  Estimation of age standardized mortality rates and gender specific cause of deaths: we will use age/sex standardized mortality estimates for comparison of study population health among study sites.
Spatiotemporal mortality by causes | 18-20 months of recruitment period
  Mapping of causes of death by location, period and seasonal variations Our field operation teams will collect the VA data with GPS installed tablets device with the purpose of assessing the location of areas with a high or low concentration of deaths in a particular time period or season.
Numbers of deaths with acute febrile illness history, to inform potential diagnostic, treatment, and referral interventions | 18-20 months of recruitment period
  Describing the number of deaths with history of fever, and/or acute febrile illnesses.
Proportion of deaths with acute febrile illness history. | 18-20 months of recruitment period
  Describing the proportion of deaths with history of fever, and/or acute febrile illnesses.
Number of causes of death reported from VA and other available sources (local treatment records, diagnoses from other SEACTN components) | 18-20 months of recruitment period
  The investigators will identify number of causes of deaths reported from VA and confirmed them against other accessible local treatment records at rural health centers or if possible, nearby hospital or findings from collected biological samples from SEACTN rural febrile illness project.

CONTACTS AND LOCATIONS:
Locations (5):
- Building Resources Across Communities (BRAC), Dhaka, Bangladesh
- villages in Thai-Myanmar border, Myawady, Kayin State, Burma
- Action for Health Development (AHEAD), Battambang, Cambodia
- Lao-Oxford-Mahosot Hospital-Wellcome Trust Research Unit (LOMWRU), Vientiane, Laos
- Chiangrai Clinical Research Unit (CCRU), Chiang Rai, Thailand